CLINICAL TRIAL: NCT04480801
Title: The Effect of Thermal Evaluation in Prevention of Diabetic Foot Ulcer: Randomized Controlled Trial
Brief Title: The Effect of Thermal Evaluation in Prevention of Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Özkal (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Sponsor-Investigator, Fatma Özkal, Lecturer, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FOzkal
Record Dates: First submitted 2020-07-02; First posted 2020-07-21 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Foot
Keywords: Diabetes Mellitus; diabetic foot; risk factors; thermal evaluation
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thermal evaluation and foot care (Experimental): Participants in the experimental group will be given foot care in the clinic and will be taught to the patient and / or their relatives. The foot care video will be uploaded to the patient and / or relative's phone. Thermal evaluation will be done. The application of the thermal evaluation, the foot areas to be applied and how to record the results of the application will be taught to the patient and / or their relatives. In addition, the thermal evaluation video will be uploaded to the phone of the patient and / or their relative. While the participants in the experimental group were discharged; Blood glucose monitoring chart, Checklist to record foot care interventions, Thermal evaluation registration form, Daily step number registration form will be provided and participants will be invited to check every 2 months.
  Interventions: Other: Thermal Evaluation and Foot Care
- foot care (Other): Participants in the control group will be given foot care in the clinic and will be taught to the patient and / or their relatives. The foot care video will be uploaded to the patient and / or relative's phone.While the participants in the control group were discharged; Blood glucose monitoring chart, Checklist to record foot care interventions will be provided and participants will be invited to check every 2 months.
  Interventions: Other: Foot Care

INTERVENTIONS:
Other: Thermal Evaluation and Foot Care — Participants in the experimental group will be given foot care and thermal evaluation in the clinic and will be taught to the patient and / or their relatives. Thermal evaluation and foot care video will be uploaded to the patient and / or relative's phone.
  Arms: thermal evaluation and foot care
Other: Foot Care — Participants in the control group will be given foot care in the clinic and will be taught to the patient and / or their relatives. Foot care video will be uploaded to the patient and / or relative's phone.
  Arms: foot care

SUMMARY:
The study was planned as a prospective randomized controlled clinical trial to determine the effect of thermal evaluation in preventing diabetic foot ulcers in patients with Type II Diabetes Mellitus (DM).

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic disease caused by insufficient production of insulin hormone in the pancreas gland or inefficient use of the insulin produced. Diabetic neuropathy that occurs in 60-70% of patients with DM is reported to be the most important factor increasing the risk of diabetic foot. Determining risk factors in diabetic foot and attempting to eliminate or mitigate these factors have been found to be a simple, inexpensive and evidence-based tool that can be used at home by patients. This study will contribute to the current literature on the effectiveness of thermal assessment in preventing diabetic foot ulcers. The study was planned as a prospective randomized controlled clinical trial to determine the effect of thermal assessment on preventing diabetic foot ulcers in patients with Type II Diabetes Mellitus (DM). For the sample of the study, compared to those with thermal evaluation, the study reported that the probability of developing diabetic feet was 10.3 times higher than those without thermal evaluation program, 48 patients (thermal evaluation group: 24 people; control group: 24 people) were included in the study. It was decided that 30 patients were lost during data collection and 35 patients were included in each study group and the study was completed with a total of 70 patients. The patients included in the study will be assigned to the experimental group (thermal evaluation group) and control group by block randomization method according to the randomization list in a ratio of 1: 1. In the study, block randomization was performed by a statistician based on the current disease year (diabetes year) and the degree of diabetic foot risk.

For the implementation of the study, permission was obtained from the ethics committee of Necmettin Erbakan University Meram Medical Faculty, Non-Drug and Medical Device Research Ethics Committee, and work permit was obtained from Necmettin Erbakan University Meram Medical Faculty Hospital Chief Physician. Patients included in the study sample will be informed before the study that the purpose of the study and participation in the study is in line with the principle of volunteering, and "Informing and Consent of Volunteers Consent Form" will be signed.

Data collection tools;

* Personal Information Form,
* Chart to Record Diabetic Foot Risk Assessment Findings
* Structured Daily Foot Care Form,
* Evaluation Charts to be Given to Patients During Discharge

Independent variables

* Identifying features of patients
* Features of patients associated with Diabetes Mellitus and its treatment
* Diabetic foot risk assessment results
* Foot care initiatives

Dependent Variables

- Development of diabetic foot ulcer

Evaluation of the Data

In the evaluation of the descriptive data obtained from the research, number, percentage, average and standard deviation will be used; The conformity of the data to normal distribution will be determined by Kolmogorov-Smirnov test and normal distribution curve, Skewness and Kurtosis test, and when the data show normal distribution, parametric tests will be used, and nonparametric tests will be used in the analysis of data that do not conform to the normal distribution. Significance will be evaluated within the confidence interval of 95%, p <0.05 will be taken.

İmplementation of the research

After vascular evaluation, neuropathy evaluation, and physical evaluation of the foot, individuals with a diagnosis of type 2 diabetes aged 18 and over will be formed the sample group. Once the sample group is determined, participants will be randomly assigned to the experimental and control groups.

Participants in the experimental group will be given foot care in the clinic and will be taught to the patient and / or their relatives. The foot care video will be uploaded to the patient and / or relative's phone. Thermal evaluation will be done. The application of the thermal evaluation, the foot areas to be applied and how to record the results of the application will be taught to the patient and / or their relatives. In addition, the thermal evaluation video will be uploaded to the phone of the patient and / or their relative. While the participants in the experimental group were discharged; Blood glucose monitoring chart, Checklist to record foot care interventions, Thermal evaluation registration form, Daily step number registration form will be provided and participants will be invited to check every 2 months.

Participants in the control group will be given foot care in the clinic and will be taught to the patient and / or their relatives. The foot care video will be uploaded to the patient and / or relative's phone.While the participants in the control group were discharged; Blood glucose monitoring chart, Checklist to record foot care interventions will be provided and participants will be invited to check every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Volunteer
* Sign the informed consent form
* Diagnosed with type II Diabetes Mellitus
* No diabetic foot ulcer
* Patients with no foot or toe amputation will be admitted.

Exclusion Criteria:

* Does not sign the informed consent form
* Without a smart phone
* Diagnosed with Type I Diabetes Mellitus,
* Patients with diabetic foot ulcers
* With ankle / arm index <0.9 and >1.30,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients developing a foot ulcer | 2 months after the first assessment
  There will be a correlation between diabetic foot development and high temperature values obtained from thermal evaluation.

SECONDARY OUTCOMES:
Changes in blood sugar values | 2-month intervals until 1-year follow-up
  Changes in blood sugar levels in both groups for 12 months every 2 months
Change in foot care practices | 2-month intervals until 1-year follow-up
  Change in foot care practices for 12 months every 2 months in both groups

CONTACTS AND LOCATIONS:
Overall Officials: FATMA ÖZKAL, Principal Investigator — Necmettin Erbakan University; Serpil YÜKSEL, Phd, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol